CLINICAL TRIAL: NCT01096043
Title: A Phase IIa, 3 Strata Dose-Defining Study Evaluating the Hemodynamic Effects, Safety and Tolerability of CXL-1020 in Patients With Systolic Heart Failure
Brief Title: A Dose-Defining Study of CXL-1020 in Patients With Systolic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Cardioxyl Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CXL-1020-02
Record Dates: First submitted 2010-03-22; First posted 2010-03-30 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2012-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; ADHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Each Strata of the study will have a placebo control. In strata A, the chance of getting active drug is 4 out of 5, in Strata B the chance of getting active drug is 3 ot of 4, and in Strata C, the chance of getting active Drug is 4 out of 5. In the event that a patient is allocated to receive placebo, the treatment may be stopped if the patient's condition fails to improve or worsens during the placebo infusion.
  Interventions: Drug: Placebo
- Strata 1 CXL-1020 (Experimental): Patients assigned to CXL-1020 in strata one will have their dose increased from the initial dose 2 times during the study period. The treatment may be stopped if the patient's condition fails to improve or worsens during the infusion.
  Interventions: Drug: Strata 1 CXL-1020
- Strata 2 CXL-1020 (Experimental): In strata 2, patients who are assigned to active treatment will receive one of up to 3 possible fixed dose levels of CXL-1020 for a period of 6 hours. The treatment may be stopped if the patient's condition fails to improve or worsens during the infusion.
  Interventions: Drug: Strata 2 CXL-1020
- Strata 3 CXL-1020 (Experimental): In strata 3, patients assigned to receive CXL-1020 will receive a fixed dose of CXL-1020 for 6 hours, and then the dose may be increased or decreased, based on the investigators assessment of the patient. The treatment may be stopped if the patient's condition fails to improve or worsens during the infusion.
  Interventions: Drug: Strata 3 CXL-1020

INTERVENTIONS:
Drug: Placebo — An infusion of an identically appearing solution of sugar water will be intravenously administered.
  Other Names: BMS-986233
  Arms: Placebo
Drug: Strata 1 CXL-1020 — Intravenous infusion of CXL-1020, up-titrated, so that 3 different dosages are administered over 6 hours
  Other Names: BMS-986233
  Arms: Strata 1 CXL-1020
Drug: Strata 2 CXL-1020 — One of 3 different dosages of CXL-1020 administered at a fixed dosage level for 6 hours.
  Other Names: BMS-986233
  Arms: Strata 2 CXL-1020
Drug: Strata 3 CXL-1020 — A fixed dose level of CXL-1020 will be administered for the initial 6 hours of treatment in Strata 3 and then dosage will be altered up or downward based on the investigators observation of the patient's condition.
  Other Names: BMS-986233
  Arms: Strata 3 CXL-1020

SUMMARY:
Study CXL-1020-02 employs is designed to further define suitable clinical dosages for CXL-1020 which will be utilized in a later Phase IIb study. The study is conducted in 3 different stages called 'strata" and evaluates the potential utility of this drug for the treatment of patents who are hospitalized with heart failure.

DETAILED DESCRIPTION:
Each of the 3 strata are described below:

Invasive Strata 1: This is a randomized, double-blinded stratum that will enroll up to 65 patients who are hospitalized with symptomatic heart failure who have indwelling PA catheters allowing invasive hemodynamic evaluation. Each patient will receive a six hour intravenous infusion of either placebo or CXL-1020.

Non-Invasive Strata 2: This is a randomized, double-blinded stratum which will enroll up to approximately 72 patients (in several cohorts with 12-24 patients each) who neither require, nor have in place, an indwelling PA catheter for hemodynamic monitoring, but meet study entrance criteria for symptoms of heart failure, (dyspnea at rest)and systolic dysfunction by specific echocardiography criteria. Monitoring of drug effects will be performed by Echocardiography.

Invasive-Strata 3: This is a randomized, double-blinded stratum that will begin after an evaluation of a substantial number of patients in Strata A and B and will enroll approximately 15-30 patients using the same general enrollment criteria as in Invasive Strata A.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for randomization, a patient MUST:

* Be a male or post menopausal or surgically sterile female requiring inpatient evaluation or treatment and be between 18 and 85 years of age
* Not require immediate emergent treatment with conventional parenteral inotropes or vasodilators
* Be receiving standard background heart failure therapies as indicated, but not receive an oral dose of a hemodynamically active treatment or diuretic within 3 hours of baseline hemodynamic assessments
* Have chronic Systolic HF due to primary/idiopathic dilated cardiomyopathy, coronary artery disease or hypertension
* For inclusion in the Non-Invasive Strata B, have a baseline (within 48 hours prior to dosing) left ventricular ejection fraction ≤ 35% estimated from a baseline 2D-Echocardiogram
* For inclusion in the Invasive Strata A and C, have baseline hemodynamic values (mean of 3 consecutive CI measurements taken within 1 hours preceding dosing within 10% of one another with a mean CI of less than or equal to (≤) 2.5L/min AND a mean PCWP of greater than 20mmHg
* Have an elevated baseline BNP of at least 400pg/ml in all protocol strata
* Be capable of understanding the nature of the trial and be willing to participate as documented by written informed consent
* Be willing and able to comply with the inpatient and outpatient study protocol requirements for the duration of the study (treatment plus 30 follow up at days)
* If a post-menopausal or surgically sterile female, confirmation of sterility status (post-menopausal or surgically sterile for at least 6 months; post-menopausal subjects will require a urine pregnancy test for confirmation)
* If a fertile male, must be using 2 approved contraceptive methods (a condom and a spermicidal agent, even if partner(s) is using birth control) for 10 days following participation in the study and further agree to not donate sperm for 10 days after participation in the study
* Must have a negative urine test for drugs of abuse and a negative ethanol breath test or blood test at baseline before dosing
* Have required local laboratory safety data within protocol required or local laboratory non-exclusionary ranges before dosing
* May be receiving ICD, Bi V pacing or rate control pacing at the time of randomization so long as no alteration of settings are anticipated within the day of study drug administration

  * Exclusion Criteria:

In order to be eligible for randomization, a patient MUST NOT:

* Have participated in any investigational drug study, SERCa gene therapy or cellular myocardial transplant study within 30 days preceding randomization or have previously received therapy with CXL-1020
* Have received a parenteral or oral dose of diuretics or other hemodynamically active therapy within 3 hours of the baseline hemodynamic assessment
* Have received intravenous inotropes, inodilators or vasodilators (amrinone, digoxin, dopamine, dobutamine, enoximone, levosimendan, milrinone, nesiritide, nitroglycerine or nitroprusside) for more than 4 hours and within 12 hours prior to randomization to treatment with study drug
* Have a heart rate <50 or ≥ 90 BPM at baseline prior to randomization
* Have a blood pressure >150 Systolic and/or >95 diastolic mmHg at baseline prior to randomization
* Have a systolic blood pressure of less than 100 mmHg at baseline prior to randomization
* Be in atrial fibrillation/flutter at the time of randomization or have a history of recent intermittent A-fib/flutter within the previous week
* Have non-sustained VT (HR > 120 bpm) of 10 beats or more during bedside monitoring prior to randomization or excessive VPB's or complex multifocal ventricular ectopy exceeding 10 beats per minute on a 2 minute rhythm strip taken within 10 minutes prior to randomization
* Have a history of successful cardiac resuscitation within the past 2 years. (Inappropriate ICD firings for non lethal arrhythmias are not exclusionary)
* Be hospitalized with acute coronary syndrome or acute myocardial infarction during the previous 90 days prior to randomization
* Have a history of stroke (CVA) or transient ischemic attack (TIA) within six months prior to randomization
* Have a concurrent history of CCS Class III or IV angina
* Be a patient whose HF etiology is attributable to either restrictive/obstructive cardiomyopathy, idiopathic hypertrophic cardiomyopathy (as defined by any wall thickness > 1.8 cm) or uncorrected severe valvular disease
* Be receiving concomitant oral or parenteral therapy with any antiarrhythmic drugs other than amiodarone or dronedarone. (only oral therapy is allowed for these agents)
* Have unsuitable echocardiographic windows for the Echo assessments (applies only to Strata B)
* Have a screening or baseline serum Na < 130 mEq/l or > 145 mEq/l; a serum K < 3.5 mEq/l or > 5.5 mEq/l; a serum Ca < 7.5 mg/dl or > 10.2 mg/dl; or a serum Mg < 1.6 mEq/l or > 3.0 mEq/l., or a digoxin level above 1ng/ml
* Have a baseline serum creatinine > 2.5 mg/dl; an ALT or AST >3 times the upper normal limit; or a hemoglobin < 10 g/dl
* Have taken ethanol within 24 hours (with a positive ethanol breath test or blood test) or a PDE5 inhibitor within 96 hours of study drug administration
* Have other clinically significant laboratory or medical conditions that, in the opinion of the Investigator, make the patient unsuitable for evaluation in the study
* Be receiving a drug which is expected to possess the potential for a clinically significant pharmacokinetic interaction with CXL-1020, as defined in the investigational drug brochure (IDB).
* Be the recipient of a myocardial restraint device or flap
* Have an anticipated survival of less than 90 days for any reason Note: Patients receiving cardiac resynchronization therapy for HF are eligible and pacemaker settings have not been changed on this hospitalization and can be left unchanged for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety and Hemodynamic Effects | At 6 Hours following start of dosing
  Define the safety and hemodynamic benefit of CXL-1020 based upon the change from baseline in hemodynamic measurements at the 6 hour time point in all strata

SECONDARY OUTCOMES:
Measurement of Plasma BNP Levels | At 6 hours following the start of dosing
  Evaluate the effects of CXL-1020 on change from baseline in circulating BNP levels after 6 hours of treatment in all strata.
Assessment of the dose/plasma concentration/effect relationship of CXL-1020 | At 6 hours following start of dosing
  Correlation of plasma concentrations of the CXL-1020 metabolites with Drug Hemodynamic Effects
Effects of CXL-1020 on Renal Function | 24 hours post dosing
  Evaluate effects of CXL-1020 on renal function parameters (serum creatinine, Cystatin C, and plasma NGAL)
Signs and Symptoms of Heart failure | At 6 hours following the start of dosing
  Evaluate heart failure symptoms in using a Likert 7-point heart failure symptom scale completed by the Investigator and a visual analogue scale completed by the patient and after the 6 hour timepoint in Stratum C
Evaluation of all Adverse Events | Through 30 days following study drug dosing
  Assess adverse events within 30 days of treatment as adjudicated by an independent safety committee (all strata)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Colucci, M.D., Study Chair — Boston University
Locations (15):
- United States (15):
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - Florida Hospital Transplant Center, Orlando, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - DMC Cardiovascular Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Medicine & Dentistry of New Jersey - New Jersey Medical School, South Orange, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Davis Heart & Lung Research Institute, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Center PA, Germantown, Tennessee

REFERENCES:
- [Derived] Sabbah HN, Tocchetti CG, Wang M, Daya S, Gupta RC, Tunin RS, Mazhari R, Takimoto E, Paolocci N, Cowart D, Colucci WS, Kass DA. Nitroxyl (HNO): A novel approach for the acute treatment of heart failure. Circ Heart Fail. 2013 Nov;6(6):1250-8. doi: 10.1161/CIRCHEARTFAILURE.113.000632. Epub 2013 Oct 9. PMID 24107588